CLINICAL TRIAL: NCT00014313
Title: A Phase II Study to Evaluate the Role of Weekly Cisplatin With Oral Etoposide in Ewing's Sarcoma and Primitive Neuroectodermal Tumor (PNET) With Bone and/or Bone Marrow Metatstatic Disease
Brief Title: Chemotherapy in Treating Patients With Metastatic Ewing's Sarcoma or Primitive Neuroectodermal Tumor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62993; EORTC-62993
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Sarcoma
Keywords: metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Cisplatin; Etoposide

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic Ewing's sarcoma or primitive neuroectodermal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of cisplatin and etoposide in terms of response of patients with metastatic Ewing's sarcoma or primitive neuroectodermal tumor.
* Assess the bone marrow and kidney toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cisplatin IV over 3 hours on days 1, 8, 15, 29, 36, and 43 and oral etoposide daily on days 1-15 and 29-43 in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 21-45 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Ewing's family tumor as characterized by the following:

  * Positive MIC2 on immunohistochemistry OR
  * Evidence of a chromosomal translocation involving the EWS gene by conventional cytogenetics

    * t(11; 22) translocation or variant OR
    * Demonstration of EWS/FLI1 or EWS/ERG gene fusion by PCR or FISH
* Metastases outside the lung or pleura
* At least 1 measurable lesion outside of previously irradiated area
* No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 15 to 65

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin less than 3 mg/dL
* Albumin greater than 2.5 g/dL

Renal:

* Creatinine less than 1.2 mg/dL
* Creatinine clearance greater than 70 mL/min

Cardiovascular:

* No history of uncontrolled cardiovascular disease

Other:

* No other severe medical illness, including psychosis
* No other prior primary malignancy except adequately treated carcinoma in situ of the cervix or basal cell skin cancer
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2001-01; Primary Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R. Judson, MA, MD, FRCP, Study Chair — Institute of Cancer Research, United Kingdom
Locations (1):
- Institute of Cancer Research - UK, Sutton, England, United Kingdom